CLINICAL TRIAL: NCT01593865
Title: Observational, Case-Control, Propensity-Matched Study of Bilateral Versus Monolateral Internal Mammary Artery Grafting for Severe Coronary Artery Disease. Assessment of Feasibility of Systematic Bilateral Mammary Artery Grafting and Early/Late Clinical Outcomes
Brief Title: The Catholic University BIMA Grafting Study
Acronym: CATHEXIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Catholic University, Italy (Other)
Responsible Party: Principal Investigator, Mario Gaudino, Researcher at Cardiac Surgery University Department, Catholic University, Italy
Other Study IDs: CathUni001
Record Dates: First submitted 2012-05-05; First posted 2012-05-08 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-08

CONDITIONS: Multivessel Coronary Artery Disease
Keywords: Coronary Artery Bypass Grafting; Mammary Artery Grafts; Bilateral Mammary Artery Grafting; Clinical Outcomes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- BIMA Grafting Group: Group consists of patients who received bilateral internal mammary artery grafting for treatment of severe coronary disease since June 2012.
  Interventions: Procedure: BIMA Grafting
- Control Group: This Group consists of historical control patients who received conventional coronary artery bypass grafting (left mammary artery graft only plus great saphenous vein grafts) in the 2010-2012 period, and who are propensity-matched to the BIMA Group patients.
  Interventions: Procedure: Left-only mammary artery grafting

INTERVENTIONS:
Procedure: BIMA Grafting — Both the left and the right internal mammary arteries are harvested and used to revascularize the two major coronary targets. Further coronary targets may be revascularized using either great saphenous vein or radial artery grafts, if present.
  Groups: BIMA Grafting Group
Procedure: Left-only mammary artery grafting — These patients had only the left mammary artery harvested and used to revascularize the major coronary target. Great saphenous vein grafts and/or radial artery grafts were employed to revascularize the remaining targets.
  Groups: Control Group

SUMMARY:
The present study hypothesizes that the systematic use of bilateral internal mammary artery (BIMA) grafting is feasible in the practice of a University Cardiac Surgery Institution for the treatment of multivessel coronary artery disease (primary hypothesis). The secondary study hypothesis is that the BIMA grafting meets the safety endpoint compared with the conventional surgical strategy entailing left mammary artery grafting plus great saphenous vein grafts to revascularize the remaining coronary targets. The tertiary study hypothesis is that the BIMA grafting yields better follow-up results in terms of recurrence of symptoms related to coronary disease, of repeat revascularization and of cardiac mortality compared with patients treated with the conventional surgical strategy entailing left mammary artery grafting plus great saphenous vein grafts to revascularize the remaining coronary targets.

ELIGIBILITY:
Inclusion Criteria:

* Patiens undergoing primary or elective-urgent isolated multivessel Coronary Artery Bypass Grafting (CABG) Surgery

Exclusion Criteria:

* Emergency status
* Previous cardiac operation
* Any associated cardiac procedure other than CABG Surgery
* Left Ventricular Ejection Fraction <20%

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target study population consists of 1,000 patients undergoing isolated coronary surgery for multivessel disease within a Cardiac Surgery University Department.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-04; Primary Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of systematic BIMA grafting | 2012-2014 (2 years)
  Starting in June 2012, all clinical data concerning patients undergoing BIMA grafting are recorded, including the baseline demographics and risk factors, the operative time, all in-hospital complications, duration of Intensive care Unit and Hospital stays, the amount of transfusion of blood products.

SECONDARY OUTCOMES:
Clinical results at follow-up | 2012-2016 (4 years)
  The patients enrolled in the study are subjected to longitudinal follow-up to determine the rate of residual myocardial ischemia (periodical stress ECG), of recurrent symptoms of coronary disease, and of any adverse cardiac event (periodical follow-up visits).

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Massetti, MD, Study Director — Division of Cardiac Surgery, Catholic University
Locations (1):
- Policlinico Universitario "A. Gemelli", Rome, Italy, Italy